CLINICAL TRIAL: NCT01870037
Title: Phase 1 Double Blind, Placebo Controlled Study Assessing Safety and Activity Of 2 Escalating Doses of hMaxi-K Gene Transfer By Direct Injection Into the Bladder Wall In Female Subjects With OAB
Brief Title: Phase 1 Study With OAB Assessing the Safety and Activity of hMaxi-K Gene Transfer
Acronym: OAB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Urovant Sciences GmbH (Industry)
Collaborators: Ion Channel Innovations (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: ION 03-OAB
Record Dates: First submitted 2013-06-03; First posted 2013-06-05 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; OAB; gene therapy
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: sequential, dose escalation
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (PBS-20% sucrose) (Placebo Comparator): PBS-20% sucrose administered during two single-treatment dose levels (16000 micrograms [µg] and 24000 µg) by direct bladder wall intramuscular injections, 20 to 30 injections depending on active dose comparator.
  Interventions: Drug: Placebo (PBS-20% sucrose)
- hMaxi-K 16000 µg (Experimental): Single treatment (16000 µg by 20 intramuscular injections). A total of 6 participants will receive hMaxi-K, and 3 will receive placebo.
  Interventions: Drug: hMaxi-K
- hMaxi-K 24000 µg (Experimental): Single treatment (24000 µg by 30 intramuscular injections). A total of 6 participants will receive hMaxi-K, and 3 will receive placebo.
  Interventions: Drug: hMaxi-K

INTERVENTIONS:
Drug: Placebo (PBS-20% sucrose)
  Other Names: Placebo
  Arms: Placebo (PBS-20% sucrose)
Drug: hMaxi-K — Single treatment/2 escalating dose levels (16000 µg and 24000 µg by intramuscular injection)
  Other Names: URO-902
  Arms: hMaxi-K 16000 µg; hMaxi-K 24000 µg

SUMMARY:
The primary objective of this study is to evaluate the safety of a single treatment of hMaxi-K compared to placebo (PBS-20% sucrose) administered by direct bladder wall injections. Two dose levels (16000 µg and 24000 µg; 20 or 30 bladder wall injections, respectively) in females with moderate Overactive Bladder/Detrusor overactivity (OAB/DO) of ≥6 months duration will be evaluated. In each dose level, 6 participants will receive hMaxi-K and 3 will receive placebo.

DETAILED DESCRIPTION:
This is a Phase 1 double-blind, placebo-controlled study assessing the safety and activity of 2 escalating doses of hMaxi-K gene transfer by direct injection into the bladder wall in female participants with OAB/DO.

The safety parameters to be monitored include: adverse events, clinical laboratory tests, electrocardiograms, and physical examinations.

The secondary objective is to evaluate the efficacy of multiple intramuscular injections of hMaxi-K compared to the control group. Efficacy parameters that will be evaluated are: number of micturitions per 24 hours, volume per micturition, incontinence episodes, pad weight measurement of accidental bladder leaks, uninhibited contractions during cystoscopy and other cystoscopic evaluations, and general and bladder-specific quality of life assessments (Kings Health Questionnaire, SF-12 Health Survey, and International Consultation on Incontinence Questionnaire [ICIQ-SF]).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women of ≥18 years of age and non-childbearing potential
2. Symptoms of overactive bladder for ≥6 months including at least one of the following:

   1. Frequent micturition ≥8 times per 24 hours
   2. Urinary urgency or nocturia
   3. Urge urinary incontinence five or more incontinence episodes per week
3. Detrusor overactivity with ≥1 uncontrolled phasic contraction(s) of the detrusor of at least 5 centimeters/H20 pressure documented on cystometry at Screening Visit 1A
4. Residual urine volume of ≤200 milliliters (ml)
5. Non-response or poor tolerance to previous treatment for symptoms of OAB/urinary incontinence and do not wish to continue these treatments
6. Have screening laboratory values and electrocardiogram that are within the normal range
7. Able to understand study requirements (i.e., literate in English), give written informed consent, and comply with all study procedures and requirements.

Exclusion Criteria:

* A woman with a positive serum (HCG) pregnancy test or who is lactating
* History of three or more culture-documented recurrent urinary tract infections per year
* Current history or previous diagnosis of painful bladder syndrome (interstitial cystitis) with pain in the region of the pelvis, perineum, or lower abdomen relieved by voiding
* Current history of neurological bladder dysfunction
* A life expectancy of less than 12 months
* Current history of Grade 2 or greater cystocele
* An indwelling urethral catheter or need for clean intermittent self-catheterization
* Recent heart attack
* Uncontrolled diabetes
* Latex allergy
* Stress urinary incontinence as determined by observation of the participant coughing while standing with a full bladder and/or response of 2 or 3 on the following Stress Urinary Incontinence question: Do you experience leakage when laughing, coughing, lifting heavy objects or other types of discreet, moderately intense activities? 0=NONE: No leakage. 1=MILD: Minimal leakage on rare occasions during these types of activities; easily tolerated; do not use pads for this. 2=MODERATE: Enough leakage that it requires occasional use of pads and may interfere with usual activity and tasks. 3=SEVERE: Extreme leakage and discomfort that stops all activity and tasks and requires the use of pads on all occasions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-02-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with any treatment-emergent adverse event during the Treatment Period | 6 months (24 weeks) per participant
Number of participants with any treatment-emergent adverse event during the Safety Follow-up Period | 18 months
Number of participants with any clinically significant clinical laboratory test value during the Treatment Period | 6 months (24 weeks) per participant
Number of participants with any clinically significant clinical laboratory test value during the Safety Follow-up Period | 18 months
Number of participants with any clinically significant electrocardiogram finding during the Treatment Period | 6 months (24 weeks) per participant
Number of participants with any clinically significant electrocardiogram finding during the Safety Follow-up Period | 18 months
Number of participants with any clinically significant physical examination finding during the Treatment Period | 6 months (24 weeks) per participant
Number of participants with any clinically significant physical examination finding during the Safety Follow-up Period | 18 months

SECONDARY OUTCOMES:
Change from Baseline in the number of micturitions per day | Baseline; 6 months (24 weeks) per participant
Change from Baseline in the volume of micturitions | Baseline; 6 months (24 weeks) per participant
Change from Baseline in incontinence episodes | Baseline; 6 months (24 weeks) per participant
Change from Baseline in pad weight | Baseline; 6 months (24 weeks) per participant
Change from Baseline in uninhibited contractions during cystoscopy | Baseline; 6 months (24 weeks) per participant
Change from Baseline in the participant rating of the Kings Health Questionnaire (KHQ) score | Baseline; 6 months (24 weeks) per participant
Change from Baseline in the International Consultation on Incontinence Questionnaire-Short Form score | Baseline; 6 months (24 weeks) per participant
Change from Baseline in the Short Form-12 (SF-12) score | Baseline; 6 months (24 weeks) per participant

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - AccuMed Research Associates, Garden City, New York
  - NYU, New York, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared

DOCUMENTS (3):
  • Study Protocol (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT01870037/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT01870037/SAP_001.pdf
  • Informed Consent Form (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT01870037/ICF_002.pdf